CLINICAL TRIAL: NCT04591990
Title: HYdrocortisone and VAsopressin in Post-REsuscitation Syndrome
Acronym: HYVAPRESS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP200033; 2020-001620-33 (EudraCT Number)
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Postresuscitation Syndrome
Keywords: intensive care; hydrocortisone; vasopressin; post-resuscitation syndrome
MeSH Terms: conditions — Diabetes Insipidus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AVP + placebo hydrocortisone (Experimental): REVERPLEG® 40 IU/2mL+ Placebo of hydrocortisone.
  Interventions: Drug: Administration of AVP; Drug: Administration of placebo hydrocortisone
- placebo AVP + hydrocortisone (Experimental): Placebo of REVERPLEG® 40 IU/2mL + Hydrocortisone 100mg UPJOHN®.
  Interventions: Drug: Administration of placebo AVP; Drug: Administration of hydrocortisone
- AVP + hydrocortisone (Experimental): REVERPLEG® 40 IU/2mL + Hydrocortisone 100mg UPJOHN®.
  Interventions: Drug: Administration of AVP; Drug: Administration of hydrocortisone
- placebo AVP + placebo hydrocortisone (Experimental): Placebo of REVERPLEG® 40 IU/2mL + placebo of hydrocortisone
  Interventions: Drug: Administration of placebo AVP; Drug: Administration of placebo hydrocortisone

INTERVENTIONS:
Drug: Administration of AVP — Administration of AVP
  Arms: AVP + hydrocortisone; AVP + placebo hydrocortisone
Drug: Administration of placebo AVP — Administration of placebo AVP
  Arms: placebo AVP + hydrocortisone; placebo AVP + placebo hydrocortisone
Drug: Administration of placebo hydrocortisone — Administration of placebo hydrocortisone
  Arms: AVP + placebo hydrocortisone; placebo AVP + placebo hydrocortisone
Drug: Administration of hydrocortisone — Administration of hydrocortisone
  Arms: AVP + hydrocortisone; placebo AVP + hydrocortisone

SUMMARY:
The primary objective is to demonstrate the superiority of arginine-vasopressin (AVP) and hydrocortisone compared with norepinephrine regarding day-30 survival and neurological recovery in post-cardiac arrest patients with hemodynamic failure.

DETAILED DESCRIPTION:
For patients successfully resuscitated who got restoration of spontaneous circulation (ROSC) after cardiopulmonary resuscitation (CPR), the course is usually marked by a post-resuscitation syndrome including multiple organ failures of various intensity and anoxic brain damage. The cardiocirculatory failure usually dominates the clinical picture, and it often leads to multiorgan failure. This hemodynamic failure is multifactorial, including at various levels vasoplegia, myocardial dysfunction, endotoxin release and adrenal dysfunction and is at least partly related to a hormonal defect that could be counteracted by hormonal supplementation. Such a substitutive opotherapy by hydrocortisone and AVP could improve hemodynamic failure and decrease overall mortality in this setting.

This trial is a superiority multicentric trial and patients will be randomized in a 1:1:1:1 ratio using an electronic CRF.

Investigational medicinal products:

- Arginin-vasopressin or AVP (REVERPLEG) The solution for infusion is prepared by diluting 40 I.U. REVERPLEG® with sodium chloride 9 mg/ml (0.9%) solution. The total volume after dilution should be 50 ml (equivalent to 0.8 I.U. AVP per ml).

AVP will be administered according to mean arterial pressure to target a 65mmHg blood pressure for max 3 days.

- HYDROCORTISONE HEMISUCCINATE Vials with lyophilisate (100mg hydrocortisone) are provided by SERB laboratory. Hydrocortisone hemisuccinate will be administered as a 50mg intravenous bolus every 6 hours after an initial dose of 100mg, for 7 consecutive days. Stop of treatment by hydrocortisone will be performed without tapering.

Comparator treatment: placebos.

17 ICU centers in France will participate to this study targetting 380 patient's enrollment in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18y)
* Cardiac arrest (in-hospital or out-of-hospital) with sustained ROSC (> 30 minutes) admitted to the ICU
* Post-resuscitation shock defined as arterial hypotension (SAP < 90 mmHg or MAP < 65 mmHg) unresponsive to adequate fluid loading, which occurred within the first 24 hours after ROSC and requiring norepinephrine/epinephrine continuous infusion at a dose greater or equal to 0.2µg/kg/min for at least 3 hours
* A maximal delay between the start of norepinephrine infusion and randomization of 9 hours
* Informed written consent of the patient or a legally authorized close relative.

Exclusion Criteria:

* Evidence for a traumatic or a neurological cause of cardiac arrest
* Shock due to uncontrolled haemorrhage
* Previously known adrenal insufficiency
* Limitation of life-sustaining therapies
* Ongoing treatment by any steroids, whatever the dose
* Ongoing extra-corporeal circulatory assistance
* Gastrointestinal bleeding in the past 6 weeks
* Pregnant or breastfeeding women
* Participation in another interventional study involving human participants or being in the exclusion period at the end of a previous study involving human participants, if applicable
* Hypersensitivity to arginin-vasopressin and to its excipients
* Hypersensitivity to hydrocortisone and to its excipients
* Legal protection (i.e. incompetence to provide consent, guardianship, curator or incarceration)
* No affiliation with the French health care system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2021-05-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Neurological outcome | at day-30
  The primary endpoint will be the good neurological outcome at day-30. This will be evaluated using the Glasgow Outcome Scale (GOS, addendum 18.5.1) dichotomized as follow: good neurological outcome for categories 4 and 5 and poor neurological outcome or death for categories 3, 2 and 1. The GOS will be obtained at day-30 from an in-hospital visit if the patient is still hospitalized or from telephone contact with patients, relatives or general practitioners.

SECONDARY OUTCOMES:
All-cause mortality | at day-30
  Vital status at day-30.
Mortality attributed to irreversible hemodynamic failure | at day-30
  Time to irreversible cardiovascular failure defined as death in pharmacologically uncontrollable hypotension (mean arterial blood pressure < 60 mmHg) despite maximal ICU care, or withdrawal of care based on same, as previously defined (Witten L, Resuscitation 2019).
Mortality attributed to neurological withdrawal of care | at day-30
  Time to neurological withdrawal of care. Withdrawal of care will be based on expectations of a poor neurological recovery based on most recent guidelines (Sandroni C, ICM 2015).
Mortality attributed to comorbid withdrawal of care | at day-30
  Time to comorbid withdrawal of care. Comorbid withdrawal of care or refusal of life-sustaining therapy based on the expectation of a poor quality of life. This may be related to a preexisting or newly discovered terminal illness or other serious medical condition (e.g. dementia or cancer).
Day-30 brain death | at day-30
  Time to brain death (according to French legislation)
mortality attributed to recurrent cardiac arrest | at day-30
  Time to recurrent cardiac arrest
Other causes | at day-30
  Proportion of patients dead from a cause not listed above.
Neurological recovery at day-30 | at day-30
  Glasgow outcome score - extended at day-30. This score will be evaluated similarly to the primary endpoint
Brain damage | at 48 hours and at 72hours
  Neuron-specific enolase (NSE) blood level measured 48 and 72 hours after CA

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume GERI, MD, PhD, Principal Investigator — Intensive Care Unit, Clinique Ambroise Paré, 92200 Neuilly sur seine; Alain CARIOU, MD, PhD, Study Director — Medical Intensive Care Unit, Cochin Hospital, APHP, 75014 Paris
Locations (14):
- France (14):
  - Intensive care unit, CHU Amiens- Picardie, Amiens
  - Intensive care unit, CHU Angers, Angers
  - Intensive care unit, CHI Robert Ballanger, Aulnay-sous-Bois
  - Medical Intensive Care Unit, Ambroise Paré hospital, APHP, Boulogne-Billancourt
  - Intensive care unit, CH public du Cotentin, Cherbourg
  - Intensive care unit, CHU Dijon, Dijon
  - Intensive care unit, Hospices civils de Lyon, Lyon
  - Intensive care unit, Hôpital Jacques Cartier, Massy
  - Intensive care unit, CHU Montpellier, Montpellier
  - Intensive care unit, Brabois hospital, Nancy
  - Intensive care unit, Hotel Dieu hospital, Nantes
  - Intensive care unit, Clinique Ambroise Paré, Neuilly-sur-Seine
  - Intensive care unit, Cochin hospital, APHP, Paris
  - Intensive care unit, André Mignot hospital, Versailles

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Witten L, Gardner R, Holmberg MJ, Wiberg S, Moskowitz A, Mehta S, Grossestreuer AV, Yankama T, Donnino MW, Berg KM. Reasons for death in patients successfully resuscitated from out-of-hospital and in-hospital cardiac arrest. Resuscitation. 2019 Mar;136:93-99. doi: 10.1016/j.resuscitation.2019.01.031. Epub 2019 Jan 30. PMID 30710595
- [Derived] Geri G, Lascarrou JB, Levy B, Asfar P, Muller G, Legriel S, Ricome S, Cour M, Klouche K, Sauneuf B, Quenot JP, Bougouin W, Cariou A; HYVAPRESS investigators. Hydrocortisone and arginine vasopressin in post-resuscitation shock: the HYVAPRESS trial. Resusc Plus. 2025 May 19;24:100982. doi: 10.1016/j.resplu.2025.100982. eCollection 2025 Jul. PMID 40503090